CLINICAL TRIAL: NCT04257318
Title: Clitoris Potential Analgesic Function Research by Pregnant Women : Feasibility Study
Acronym: FAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2018/0415/HP
Record Dates: First submitted 2020-01-29; First posted 2020-02-06 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Pregnancy Related

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vibrating Relaxation Tool (Experimental): Use of a Vibrating Relaxation Tool in case of pain during pregn
  Interventions: Other: Vibrating Relaxation Tool

INTERVENTIONS:
Other: Vibrating Relaxation Tool — Use of a Vibrating Relaxation Tool in case of pain during pregnancy

SUMMARY:
Assessment of the acceptability by pregnant women on the research of the potential analgesic function of the clitoris.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman, whatever the term, primiparous or multiparous
* Age ≥ 18 years old
* Patient having read and understood the information letter and signed the consent form
* Patient affiliated to Social Security

Exclusion Criteria:

* Inability to understand French or information,
* Person deprived of their liberty by an administrative or judicial decision
* Person placed under the protection of justice
* Person under guardianship or curatorship

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-08-11 (Actual); Primary Completion 2022-11-02 (Actual); Study Completion 2022-11-02 (Actual)

PRIMARY OUTCOMES:
Acceptability | through study completion, an average of 15 months
  Among patients who had the information visit, proportion of those who were included and applied the procedure at least twice

CONTACTS AND LOCATIONS:
Overall Officials: Eric VERSPYCK, Pr, Principal Investigator — University Hospital, Rouen; Manon BESTAUX, Dr, Principal Investigator — University Hospital, Rouen
Locations (1):
- Rouen University Hospital, Rouen, France